CLINICAL TRIAL: NCT00955539
Title: The Importance of Viability for Response to Cardiac Resynchronization Therapy
Brief Title: Viability and Cardiac Resynchronization Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Lund University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Risum, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-B-2009-057
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy
Keywords: Heart Failure; Cardiac resynchronization therapy; Optimization; Viability; Mechanical dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT group 1 (Active Comparator)
  Interventions: Device: AV-optimization followed by AV- and VV-optimization
- CRT group 2 (Active Comparator)
  Interventions: Device: AV- and VV-optimization followed by AV-optimization only.

INTERVENTIONS:
Device: AV-optimization followed by AV- and VV-optimization — Patients are AV-optimized the first 4 months,then AV- and VV-optimized the next 4 months.
  Arms: CRT group 1
Device: AV- and VV-optimization followed by AV-optimization only. — Patients are AV- and VV-optimized the first 4 months,then AV-optimized the next 4 months.
  Arms: CRT group 2

SUMMARY:
30% of heart failure patients that receive a device for cardiac resynchronization therapy fail to show clinical improvement. The reason for lack of response is still unclear but factors such as scar tissue in the heart musculature, inadequate lead placement, device-settings and the degree of dyssynchrony before implant seems to be important. In this study, these factors are further investigated.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is an established therapy for patients with severe heart failure, depressed left ventricular function and a wide QRS-complex. Large clinical trials have demonstrated unequivocal improvements in functional status, morbidity and mortality. However, 30 % of heart failure patients treated with a CRT-device do not benefit clinically. Several factors have been suggested to be important for the response to CRT such as mechanical dyssynchrony, presence of scar tissue in the myocardium, and device-optimization (among others). It is the purpose of this study to investigate the importance of these factors.

100 patients with ischemic cardiomyopathy, eligible to CRT according to current guidelines, will be included. Patients are randomised to two arms. One group will have atrioventricular (AV)-optimization after implantation, the other AV -and interventricular (VV)-optimization. After 4 months patients are crossed-over to the other arm. Preimplantation patients are MR-scanned and low-dose dobutamine stress-echocardiography is performed. Furthermore patients will be examined by echocardiography and evaluation of clinical status

1. Mechanical dyssynchrony can predict response to CRT. b. Measures of mechanical dyssynchrony is related to myocardial viability and conduction.
2. Individual optimization based on conduction times will increase benefit to CRT. b. The effect of adding VV-optimization is related to myocardial viability.
3. > 30 % of non-viable tissue globally in the myocardium is predictive of lack of CRT- response. b. Non-viable tissue located in the area of the left ventricular lead is predictive of non-response.

ELIGIBILITY:
Inclusion Criteria:

* LVEF</= 35%, QRS-duration>/= 120 ms, NYHA-class II- IV.
* Ischemic heart disease (> 50% stenosis in 1 or more major epicardial coronary artery or prior PCI or CABG.)
* Optimal treatment ( beta-blocker, ACE-1 or ARB and spironolactone)

Exclusion Criteria:

* Pregnancy
* Unstable angina pectoris
* Chronical atrial fibrillation
* Severe valvular disease
* Dementia or mental retardation
* Severe claustrophobia
* Acute myocardial infarction < 3 months
* Severe health condition threatening short-term survival
* Severe kidney insufficiency, GFR < 35 ml/min/1.73 m2
* Metal implants contraindicative of magnetic resonance scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Responders:Echocardiographic:>/= 10% increase in Left ventricular ejection fraction (LVEF) or >/= 15 % reduction in left ventricular end-systolic volume (LVESV) | 4 and 8 months, ( follow up- 2 years)

SECONDARY OUTCOMES:
LVESV, LVEDV, Cardiac output (CO), Minnesota Living with Heart Failure Questionnaire (MLHFQ) ProBNP Others: t-wave modulation all-cause mortality, cardiac death, hospitalization | 4 and 8 months (follow-up after 2 years)
Clinical: >/= 25% increase in 6-min walk test or >/= 1 reduction in NYHA-class | 4 and 8 months (follow-up 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Risum, M.D., Principal Investigator — University Hospital Gentofte, Department of cardiology; Thomas Fritz Hansen, M.D., Study Chair — University Hospital Gentofte, department of cardiology; Peter Søgaard, M.D., DMSc., Study Chair — Gentofte University Hospital, department of cardiology; Rasmus Borgquist, MD, PhD, Study Chair — University Hospital Lund; Niels E Bruun, MD, DMSc, Study Chair — Gentofte University Hospital, department of cardiology
Locations (2):
- Gentofte University Hospital, Hellerup, Denmark
- University Hospital Lund, Lund, Lund, Sweden

REFERENCES:
- [Background] Bax JJ, Abraham T, Barold SS, Breithardt OA, Fung JW, Garrigue S, Gorcsan J 3rd, Hayes DL, Kass DA, Knuuti J, Leclercq C, Linde C, Mark DB, Monaghan MJ, Nihoyannopoulos P, Schalij MJ, Stellbrink C, Yu CM. Cardiac resynchronization therapy: Part 1--issues before device implantation. J Am Coll Cardiol. 2005 Dec 20;46(12):2153-67. doi: 10.1016/j.jacc.2005.09.019. PMID 16360042
- [Background] Sogaard P, Egeblad H, Pedersen AK, Kim WY, Kristensen BO, Hansen PS, Mortensen PT. Sequential versus simultaneous biventricular resynchronization for severe heart failure: evaluation by tissue Doppler imaging. Circulation. 2002 Oct 15;106(16):2078-84. doi: 10.1161/01.cir.0000034512.90874.8e. PMID 12379577
- [Background] Bleeker GB, Kaandorp TA, Lamb HJ, Boersma E, Steendijk P, de Roos A, van der Wall EE, Schalij MJ, Bax JJ. Effect of posterolateral scar tissue on clinical and echocardiographic improvement after cardiac resynchronization therapy. Circulation. 2006 Feb 21;113(7):969-76. doi: 10.1161/CIRCULATIONAHA.105.543678. Epub 2006 Feb 13. PMID 16476852
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115